CLINICAL TRIAL: NCT01202786
Title: An Exploratory Cost-effectiveness Study of miRview™ Mets in Patients With Cancer of Unknown Primary (CUP) in Israel
Brief Title: Cost-effectiveness Study of miRview™ Mets in Patients With Cancer of Unknown Primary (CUP)
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Clalit Health Services (Other); Rosetta Genomics (Unknown)
Responsible Party: Sponsor
Other Study IDs: ONCO1miRviewmets
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Neoplasms, Unknown Primary
Keywords: Cancer of Unknown Primary Site (CUP)
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin Fixed Paraffin Embedded tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- miRview mets Disclosed: Patients of group 1 will be submitted to the standard conventional work-up (see below) as well as miRview™ mets assay. Their physician will treat the patient based upon both results
- Control: Patients of group 2 will be submitted to the standard conventional work-up. miRview™ mets assay will be performed but will remain blinded for both the patient and referring physician. Treatment will be decided based on standard work-up results

SUMMARY:
The aim of the study is in cancer of unknown primary (CUP) patients, to compare the cost-effectiveness of miRview™ mets test with conventional work-up in identifying the primary tumor site.

DETAILED DESCRIPTION:
Thousands of patients are diagnosed each year with metastatic cancer; however, about 3-5% of them are diagnosed with Cancer of Unknown Primary (CUP). In order to identify the optimal treatment plan for individual patients with CUP, the primary tumor site must be identified. Patients undergo a wide range of costly, time-consuming, and inefficient tests to identify the primary site of origin, often to no avail.

In this era of targeted therapies, the accurate diagnosis of the primary tumor can be crucial. miRview™ mets is a new molecular diagnostic tool that identifies the tissue-of-origin of metastatic tumors, with 90% sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who present with histologically-confirmed metastatic cancer in whom an initial work-up which consists of detailed medical history, physical examination, basic laboratory studies, histopathological review of biopsy material, and CT scan of the chest abdomen and pelvis fail to identify the primary site.
2. Older than 18 years
3. Performance status <2
4. life expectancy >3 months
5. ANC >1500
6. Platelets >100,000 if bone marrow is not involved
7. Hb > 9
8. Creatinine <2
9. LFTS < x5 normal
10. Histology proven of malignancy
11. Enough material for miRview test (10 slices of 10 micrometer sections)
12. Member of Clalit HMO

Exclusion Criteria:

1. Patients unable or unwilling to sign the informed consent form
2. Under 18 years old
3. Performance status >2
4. life expectancy<3 months
5. ANC <1500
6. Platelets <100,000 if marrow not involved
7. Hb < 9
8. Creatinine >2
9. LFTS > x5 normal
10. Not member of Clalit HMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with histologically-confirmed metastatic cancer in whom an initial work-up which consists of detailed medical history, physical examination, basic laboratory studies, histopathological review of biopsy material, and CT scan of the chest abdomen and pelvis fail to identify the primary site.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
cost-effectiveness | 18 months
  To compare the cost-effectiveness of miRview™ mets test with conventional work-up in cancer of unknown primary (CUP) patients, by comparing total cost and time of the diagnostic process (including hospitalization time) from day 1 of the study to the decision on treatment program

SECONDARY OUTCOMES:
compare the diagnostic performance | 18 months
  1. Evaluating the miRview™ mets results based on the clinical and pathological work-up in all patients (retrospectively).
  2. Evaluating the concordance between miRview™ mets result and the diagnosis obtained by the standard work-up process.
  3. Comparing the response to treatment between study groups.
  4. Comparing overall survival between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Salomon Shtemmer, MD, Principal Investigator — Clalit Health Services
Locations (3):
- Israel (3):
  - Ha'emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rabin Medical Center, Petah Tikva